CLINICAL TRIAL: NCT00341705
Title: The Second Multicenter Hemophilia Cohort Study
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Multicenter Hemophilia Cohort Study (Unknown)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999901170; 01-C-N170
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2013-04-02

CONDITIONS: Liver Decompensation; Hepatocellular Carcinoma; Non-Hodgkin Lymphoma
Keywords: AIDS; Cancer; Hepatitis C Virus; HIV; Natural History; Hemophilia; Hepatitis C
MeSH Terms: conditions — Hepatic Insufficiency; Carcinoma, Hepatocellular; Lymphoma, Non-Hodgkin; Acquired Immunodeficiency Syndrome; Neoplasms; Hepatitis C; Hemophilia A

SUMMARY:
The Second Multicenter Hemophilia Cohort Study (MHCS-II) will evaluate and prospectively follow approximately 4500 persons with hemophilia who were exposed to hepatitis C virus (HCV). The vast majority will have been infected with HCV, and approximately 1/3 will have been infected with human immunodeficiency virus (HIV). Primary objectives are to quantify the rates of liver decompensation, hepatocellular carcinoma, and non-Hodgkin lymphoma and to evaluate candidate clinical, genetic, virologic, serologic and immunologic markers that are likely to be on the causal pathway for these conditions. Candidate clinical and laboratory markers will be examined longitudinally to define changes over time and their relationships to one another. Collaborative studies will focus on genome scanning and evaluation of candidate genetic loci for susceptibility or resistance to HCV and HIV infections or to the diseases that result from these infections. Additional studies will identify response and complication rates of various anti-HCV and anti-HIV regimens in the setting of comprehensive clinical care of persons with hemophilia.

DETAILED DESCRIPTION:
The Second Multicenter Hemophilia Cohort Study (MHCS-II) will evaluate and prospectively follow approximately 4500 persons with hemophilia who were exposed to hepatitis C virus (HCV). The vast majority will have been infected with HCV, and approximately 1/3 will have been infected with human immunodeficiency virus (HIV). Primary objectives are to quantify the rates of liver decompensation, hepatocellular carcinoma, and non-Hodgkin lymphoma and to evaluate candidate clinical, genetic, virologic, serologic and immunologic markers that are likely to be on the causal pathway for these conditions. Candidate clinical and laboratory markers will be examined longitudinally to define changes over time and their relationships to one another. Collaborative studies will focus on genome scanning and evaluation of candidate genetic loci for susceptibility or resistance to HCV and HIV infections or to the diseases that result from these infections. Additional studies will identify response and complication rates of various anti-HCV and anti-HIV regimens in the setting of comprehensive clinical care of persons with hemophilia.

ELIGIBILITY:
* INCLUSION CRITERIA:

Must be registered patient with an inherited coagulation disorder at a participating MHCS-II center. Disorders include hemophilia A or B (congenital factor VIII or IX deficiency), deficiencies in other factors such as V or XI, and vonWillebrand's disease. (Unless noted otherwise, all of the disorders will collectively be referred to as hemophilia .) All such hemophilia and vonWillebrand s disease patients are to be recruited as study participants.

Since January 1, 1993, must have had at least one positive result on a licensed assay for HCV antibodies, HIV antibodies, or HIV RNA.

Must be at least 13 years of age at enrollment.

Must provide signed informed consent or, for minors, signed assent plus signed informed consent from the parent or guardian.

EXCLUSION CRITERIA:

Is not a patient with an inherited coagulation disorder.

Does not have a positive test for HCV antibodies, HIV antibodies, or HIV RNA on a licensed assay performed since January 1, 1993.

Is less than 13 years of age.

Lacks informed consent/assent.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2565 (Actual)
Dates: Start 2001-04-27; Study Completion 2013-04-02

CONTACTS AND LOCATIONS:
Overall Officials: James J Goedert, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (48):
- United States (39):
  - University of Arizona, Tucson, Arizona
  - University of California, Davis, Davis, California
  - Children's Hospital of Orange County, Orange, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado, Denver, Colorado
  - Christiana Hospital, Wilmington, Delaware
  - Georgetown University, Washington D.C., District of Columbia
  - Childrens National Medical Center, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - University of Illinois, Chicago, Illinois
  - Childrens Memorial Hospital, Chicago, Chicago, Illinois
  - St. Vincent's Hospital, Indianapolis, Indiana
  - Tulane University, New Orleans, Louisiana
  - Wayne State University Hutzel Hospital, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - University of Mississippi, Jackson, Mississippi
  - St. Louis University, St Louis, Missouri
  - University of New Mexico, Albuquerque, New Mexico
  - University of Buffalo, Buffalo, New York
  - North Shore Long Island Jewish Health System, Lake Success, New York
  - Cornell University, New York, New York
  - Mt. Sinai Medical Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Childrens Hospital, Cinncinati, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - Wright State University, Dayton, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Milton Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Palmentto Health Alliance, Columbia, South Carolina
  - University of Tennessee, Memphis, Tennessee
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas, Houston, Houston, Texas
  - University of Texas, San Antonio, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - Childrens Hospital of Wisconsin, Milwaukee, Wisconsin
- Brazil (2):
  - Hospital Brigadeiro, São Paulo
  - University of Sao Paulo, São Paulo
- South East Health Care Corporation, New Brunswick, Canada
- Hospices Civils de Lyon, Lyon, France
- University of Bonn, Bonn, Germany
- Laikon General Hospital of Athens, Athens, Greece
- Italy (2):
  - University of Florence, Florence
  - University de Milano, Milan
- Karolinska Institute St. Gorans Hospital, Stockholm, Sweden

REFERENCES:
- [Background] Mannucci PM, Tuddenbam EG. The hemophilias: progress and problems. Semin Hematol. 1999 Oct;36(4 Suppl 7):104-17. PMID 10595759
- [Background] Kroner BL, Rosenberg PS, Aledort LM, Alvord WG, Goedert JJ. HIV-1 infection incidence among persons with hemophilia in the United States and western Europe, 1978-1990. Multicenter Hemophilia Cohort Study. J Acquir Immune Defic Syndr (1988). 1994 Mar;7(3):279-86. PMID 8106967
- [Background] Eyster ME, Diamondstone LS, Lien JM, Ehmann WC, Quan S, Goedert JJ. Natural history of hepatitis C virus infection in multitransfused hemophiliacs: effect of coinfection with human immunodeficiency virus. The Multicenter Hemophilia Cohort Study. J Acquir Immune Defic Syndr (1988). 1993 Jun;6(6):602-10. PMID 8098752